CLINICAL TRIAL: NCT00962871
Title: An Open-label, Randomized Study to Evaluate the Acute Immunologic Responses in Asian Subjects With E Antigen Positive Chronic Hepatitis B Following Initiation of Therapy for Hepatitis B With Pegasys, Nucleoside Analogues, or Both.
Brief Title: A Study of Early Immunologic Response in Asian Patients With Chronic Hepatitis B, Treated With Pegasys (Peginterferon Alfa-2a (40KD)), Nucleoside Analogues, or Both
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP22512
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; Tenofovir

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: tenofovir
- 2 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: tenofovir
- 3 (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]
- 4 (No Intervention)

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 360 micrograms sc/week for 2 weeks
  Arms: 2; 3
Drug: tenofovir — 300mg po daily for 2 weeks
  Arms: 1; 2

SUMMARY:
This open-label, randomized, parallel-arm study will assess the early immunologic response in treatment-naïve Asian male patients with chronic hepatitis B after initiation of treatment with Pegasys or tenofovir or Pegasys plus tenofovir. Patients will be randomized to one of 4 cohorts to receive either Pegasys (360mcg subcutaneously weekly) or tenofovir (300mg orally daily) or both or no treatment for 2 weeks. After 2 weeks on study treatment, patients may opt to receive standard of care treatment with Pegasys. Target sample size is <50.

ELIGIBILITY:
Inclusion Criteria:

* male adults of Southeast and/or East Asian origin, 18-55 years of age
* HBeAg-positive chronic hepatitis B
* detectable HBV DNA

Exclusion Criteria:

* prior antiviral therapy for chronic hepatitis B
* evidence of bridging fibrosis, cirrhosis or decompensated liver disease
* positive test at screening for HAV (IgM), HCV, HDV or HIV
* history or evidence of medical condition associated with chronic liver disease
* antineoplastic or immunomodulatory treatment </=6 months prior to first dose of study drug

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (2):
  - Los Angeles, California
  - San Francisco, California
- Grafton, New Zealand
- Singapore, Singapore
- Taipei, Taiwan

REFERENCES:
- [Derived] Mehrotra A, D'Angelo JA, Romney-Vanterpool A, Chu T, Bertoletti A, Janssen HLA, Gehring AJ. IFN-alpha Suppresses Myeloid Cytokine Production, Impairing IL-12 Production and the Ability to Support T-Cell Proliferation. J Infect Dis. 2020 Jun 16;222(1):148-157. doi: 10.1093/infdis/jiaa064. PMID 32049318
- [Derived] Hong LZ, Hong S, Wong HT, Aw PP, Cheng Y, Wilm A, de Sessions PF, Lim SG, Nagarajan N, Hibberd ML, Quake SR, Burkholder WF. BAsE-Seq: a method for obtaining long viral haplotypes from short sequence reads. Genome Biol. 2014;15(11):517. doi: 10.1186/PREACCEPT-6768001251451949. PMID 25406369
- See also: This report describes the early effects of IFNα treatment on immune and viral biomarkers in HBeAg+ CHB patients. The results show that PegIFNα-induced innate immune activation directly benefits from the suppression of HBV replication. — http://www.ncbi.nlm.nih.gov/pubmed/23994382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 30 July 2009 to 01 February 2012 and recruited participants from 4 centers in New Zealand (1), Taiwan (1), and Singapore (2).
Pre-assignment Details: A total of 65 participants were screened of which 30 participants were randomized. 35 participants failed the screening evaluation mainly due to inability to meet the inclusion criteria and consent withdrawal.
Groups:
- Tenofovir 300 mg: Each participant received Tenofovir 300 mg once a day for 2 weeks and thereafter received an optional treatment of Peginterferon alfa-2a (PEG-IFN alfa-2a) 180 µg after 2 weeks of initial treatment.
- Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg: Each participant received Tenofovir 300 mg once a day and Peginterferon alfa-2a (PEG-IFN alfa-2a), 360 micrograms (µg) subcutaneously once a week for 2 weeks and thereafter received an optional treatment of Peginterferon alfa-2a (PEG-IFN alfa-2a) 180 µg after 2 weeks of initial treatment.
- PEG-IFN Alfa-2a 360 μg: Each participant received Peginterferon alfa-2a, 360 µg subcutaneously once a week for 2 weeks and thereafter received an optional treatment of Peginterferon alfa-2a (PEG-IFN alfa-2a) 180 µg after 2 weeks of initial treatment.
- Delayed Treatment: Each participant received PEG-IFN alfa-2a, 360 μg/week after an initial 2-week delay.
Period: Overall Study
Arm/Group | Tenofovir 300 mg | Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg | PEG-IFN Alfa-2a 360 μg | Delayed Treatment
Started | 6 | 6 | 12 | 6
Completed | 6 | 6 | 12 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir 300 mg | Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg | PEG-IFN Alfa-2a 360 μg | Delayed Treatment | Total
Number analyzed (Participants) | 6 | 6 | 12 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12 | 6 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.09) | 28 (3.16) | 28.5 (5.40) | 27.2 (3.87) | 30 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 12 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Viral Quantitative e Antibody
Description: An acute virologic response was determined by change from baseline in viral antigen/antibody laboratory data.
Time Frame: Day 1, 3, 5, 8, 10, 14, Week 3, 4, 5, 6 (weeks are computed from the first dose of Pegasys)
Population: All participants who received at least 1 dose of the study medication were included in this analysis. Only participants with both a baseline value and a value particular time point were summarized.
Measure: Mean (Standard Deviation); unit: Cut-off index (C.O.I.)
Arm/Group | Tenofovir 300 mg | Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg | PEG-IFN Alfa-2a 360 μg | Delayed Treatment
Number analyzed (Participants) | 6 | 6 | 12 | 6
Cut-off index (C.O.I.)
  Day 1 | 0.07 (0.162) | 0.15 (0.234) | 0.02 (0.063) | 0.03 (0.062)
  Day 3 | 0.00 (0.089) | 0.03 (0.267) | -0.13 (0.119) | -0.10 (0.274)
  Day 5 | -0.02 (0.049) | 0.04 (0.255) | -0.15 (0.150) | 0.07 (0.066)
  Day 8 | -0.05 (0.051) | 0.07 (0.223) | -0.09 (0.155) | 0.04 (0.069)
  Day 10 | -0.13 (0.146) | 0.04 (0.247) | -0.12 (0.175) | 0.03 (0.127)
  Day 14 | -0.02 (0.147) | 0.03 (0.259) | -0.13 (0.267) | -0.00 (0.162)
  Week 3 | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized | 0.01 (0.219) | -0.22 (0.282) | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized
  Week 4 | -0.04 (0.302) | -0.05 (0.370) | -0.29 (0.322) | -0.40 (0.521)
  Week 6 | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized | -0.21 (0.785) | -0.31 (0.481) | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized

2. Secondary Outcome: Mean Change From Baseline in HBV-DNA log10
Description: An acute virologic response was determined by change from baseline in HBV-DNA log10.
Time Frame: Day 1, 3, 5, 8, 10, 14, Week 3, 4, 5, 6 (weeks are computed from the first dose of Pegasys)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Tenofovir 300 mg | Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg | PEG-IFN Alfa-2a 360 μg | Delayed Treatment
Number analyzed (Participants) | 6 | 6 | 12 | 6
IU/mL
  Day 2 | -0.61 (0.330) | -0.46 (0.196) | -0.14 (0.179) | 0.08 (0.110)
  Day 3 | -1.04 (0.342) | -0.75 (0.480) | -0.46 (0.222) | 0.04 (0.064)
  Day 5 | -1.53 (0.306) | -1.45 (0.551) | -0.64 (0.239) | -0.06 (0.120)
  Day 8 | -2.16 (0.244) | -1.93 (0.645) | -0.54 (0.226) | -0.07 (0.316)
  Day 10 | -2.37 (0.167) | -2.11 (0.735) | -0.57 (0.299) | -0.09 (0.493)
  Day 14 | -2.7 (0.142) | -2.46 (0.800) | -0.61 (0.521) | -0.26 (0.573)
  Week 3 | -0.76 (0.518) | -2.88 (0.702) | -0.79 (0.622) | -1.80 (0.866)
  Week 4 | -0.84 (0.422) | -1.49 (0.652) | -0.98 (0.772) | -2.17 (0.871)
  Week 5 | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized | -1.37 (0.923) | -1.22 (0.819) | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized
  Week 6 | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized | -1.73 (1.462) | -1.30 (0.978) | NA (NA) — Only participants with both a baseline value and a value particular time point were summarized

3. Secondary Outcome: Early Changes in Viral Sequence Associated With Viral Suppression
Description: Viral sequence data was obtained from the first 10 participants enrolled in Study but on analysis of the data, numerous low frequency deviations from the HBV consensus sequences were observed in the 454 SLX sequence data which were not replicated in data obtained from routine Sanger sequencing. These sequence deviations did not correspond to a temporal pattern consistent with selection of mutations following HBV treatment. Moreover, they could not be reliably distinguished from sequencing artifacts. It was also revealed that complete genome coverage was not obtained due to errors in the design of the primer sequences. For these reasons, further sequence analyses were not performed for the remaining treatment population.
Time Frame: Day 1, 5, 14, Week 4 and 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to Week 6
Description: All participants who received at least one dose of the study medication were included in safety analysis.
Arm/Group | Tenofovir 300 mg | Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg | PEG-IFN Alfa-2a 360 μg | Delayed Treatment
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 12/12 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir 300 mg (N=6) | Tenofovir 300 mg + PEG-IFN Alfa-2a 360 μg (N=6) | PEG-IFN Alfa-2a 360 μg (N=12) | Delayed Treatment (N=6)
Pyrexia (General disorders) | 0 | 5 | 9 | 3
Fatigue (General disorders) | 2 | 2 | 4 | 2
Influenza like illness (General disorders) | 1 | 0 | 1 | 1
Pain (General disorders) | 1 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 2 | 0
Feeling cold (General disorders) | 1 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1
Xerosis (General disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 5 | 6 | 4
Lethargy (Nervous system disorders) | 1 | 1 | 3 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Wolff-parkinson-white syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.